CLINICAL TRIAL: NCT01453686
Title: A Randomized Controlled Trial of Clobetasol Propionate 0.05% Cream Versus Hydrocortisone 1% Cream in Children With Alopecia Areata
Brief Title: A Trial of Clobetasol Propionate Versus Hydrocortisone in Children With Alopecia Areata
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Patricia Parkin, Staff Paediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0020020248
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Hydrocortisone; Clobetasol Propionate; Randomized Controlled Trial
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone 1% (Experimental)
  Interventions: Drug: Hydrocortisone 1%
- Clobetasol Propionate 0.05% (Experimental)
  Interventions: Drug: Clobetasol Propionate 0.05%

INTERVENTIONS:
Drug: Hydrocortisone 1% — Topical cream, used twice daily for 6 weeks on affected area, followed by 6 weeks of no treatment, followed by an additional 6 weeks of the same intervention.
  Arms: Hydrocortisone 1%
Drug: Clobetasol Propionate 0.05% — Topical cream, used twice daily for 6 weeks on affected area, followed by 6 weeks of no treatment, followed by an additional 6 weeks of the same intervention.
  Arms: Clobetasol Propionate 0.05%

SUMMARY:
The use of topical steroids in the treatment of alopecia areata in children is common practice. However, no particular potency of steroid is accepted as the standard treatment due to the paucity of high quality evidence in the dermatology literature to substantiate their use. Two randomized controlled trials exist assessing topical steroid efficacy in this disorder, both have methodological limitations. The question remains as to which topical steroid is safe and efficacious for use. We performed a double blinded controlled trial to assess the usefulness of a class 1 topical steroid (clobestasol proprionate 0.05%) compared with a class 7 topical steroid (hydrocortisone 1%) in children with alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 16 years
* New patients presenting to The Hospital for Sick Children
* Clinical confirmation of alopecia areata
* Hair loss between 10 -75%

Exclusion Criteria:

* Skin or medical problems requiring use of oral steroids
* Immunosuppressants or PUVA for 4 weeks prior to the study
* Use of inhaled and or intranasal steroids for 14 days prior to trial
* Topical medicaments for 7 days prior to the trial

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2002-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in scalp surface area affected over time | 24 weeks
  The change in scalp surface area affected will be compared between the two intervention groups from baseline to 6 weeks, 12 weeks, and 24 weeks.

SECONDARY OUTCOMES:
Change in scalp surface area affected from baseline to end of study | 24 weeks
  The percent change in scalp surface area affected on the scalp will be compared between the intervention groups from baseline to 24 weeks.
Over 50% reduction in scalp surface area affected | 24 weeks
  The number of subjects who had over 50% reduction in scalp surface area affected from baseline to 24 weeks will be compared between the intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Macarthur, MBChB, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lenane P, Macarthur C, Parkin PC, Krafchik B, DeGroot J, Khambalia A, Pope E. Clobetasol propionate, 0.05%, vs hydrocortisone, 1%, for alopecia areata in children: a randomized clinical trial. JAMA Dermatol. 2014 Jan;150(1):47-50. doi: 10.1001/jamadermatol.2013.5764. PMID 24226568